CLINICAL TRIAL: NCT05196919
Title: A Placebo-controlled, Double-blind Evaluation of Safety, Tolerability, and Efficacy of XT- 150 for the Treatment of Facet Joint Osteoarthritis Pain
Brief Title: Safety and Efficacy of XT-150 for Facet Joint Osteoarthritis Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xalud Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XT-150-1-0302
Record Dates: First submitted 2021-12-13; First posted 2022-01-19 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Facet Joint Pain; Back Pain; Inflammation
Keywords: FJOA; Facetogenic Pain; Intra-articular Injection
MeSH Terms: conditions — Back Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled, double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.15mg XT-150 (Experimental): 0.15mg XT-150 administered in 1.0 mL total delivered by two 0.5 mL injections on Day 0 and Day 90.
  Interventions: Biological: XT-150
- 0.45mg XT-150 (Experimental): 0.45mg XT-150 administered in 1.0 mL total delivered by two 0.5 mL injections on Day 0 and Day 90.
  Interventions: Biological: XT-150
- Placebo (Placebo Comparator): Placebo administered in 1.0 mL total delivered by two 0.5 mL injections on Day 0 and Day 90.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: XT-150 — XT-150 is a plasmid Deoxyribonucleic acid (DNA) formulated in buffered, D mannose saline solution.
  Arms: 0.15mg XT-150; 0.45mg XT-150
Biological: Placebo — Phosphate-buffered saline for injection
  Arms: Placebo

SUMMARY:
This is a Phase 2a safety and efficacy study of XT-150 in adult participants experiencing back pain due to inflammation of the facet joint, also known as facet joint osteoarthritis (FJOA), and who are eligible for intra articular glucocorticoid injection, or radiofrequency ablation of medial branches of the primary dorsal ramus of the exiting nerve root, which innervates the adjacent facet joints.

Study drug will be administered at Day 0 and Day 90 by bilateral intra-articular (IA) injection into the facet capsule, at the affected spinal level (e.g. Lumbar [L]3-4, L4-5, or L5-Sacrum [S]1) as determined by imaging (e.g., Magnetic resonance imaging [MRI], Computed tomography [CT]), X-ray, etc.) and physical exam.

Up to 72 participants will be randomized to placebo or one of two dose treatment groups (24 participants per treatment group).

1. 0.15 mg XT-150 (1.0 milliliter [mL] total delivered by two 0.5 mL injections)
2. 0.45 mg XT-150 (1.0 mL total delivered by two 0.5 mL injections)
3. Placebo (Sterile saline) (1.0 mL total delivered by two 0.5 mL injections)

ELIGIBILITY:
Inclusion Criteria:

Participants are required to meet ALL of the following inclusion criteria:

1. Male or female, between 18 and 90 years of age, inclusive.
2. Sufficiently severe facet arthropathy of lumbar facets as determined by imaging (e.g., MRI, CT, X-ray, etc.) to establish an underlying basis of disease, as determined by usual bony and ligamentous signs of osteoarthritis (OA). Use of historical images permitted if obtained within the last 12 months.
3. Complaint of nociceptive, mechanical pain of lumbar spine, in particular pain localized to paramedian axis as opposed to midline or radicular. Radicular pain as a secondary finding may be allowed if it is in addition to mechanical pain and can be clinically distinguished by participant.
4. LBP (Low Back Pain) worsened by activity or motion of region
5. Have had a positive diagnostic facet pain block with lidocaine; admittance if participant gains 50% relief of pain within 30 minutes of test injection
6. Be free of local or intra-articular infection, tumor or other causes of localized LBP, for example, spondylolysis/pars defect, and adjacent vertebral body compression fracture based on imaging evaluation.
7. Symptomatic disease because of osteoarthritis, established by imaging of facet joint and defined as a worst pain of at least 50 at the Screening Visit and the Baseline (Day 0) Visit (based on scale of 0 to 100, with 100 representing "pain as bad as you can imagine") using Visual Analog Scale (VAS).
8. Stable analgesic regimen during the 4 weeks prior to enrollment. Participants who are not currently on any analgesics at the time of enrollment because they have discontinued prior analgesic therapy due to intolerance or lack of effect may be included. New analgesics or changes to the pre-established regimen during the study, with the exception of rescue medication use, are not permitted.
9. Inadequate pain relief with prior therapies lasting 3 months or more.
10. In the judgment of the Investigator, acceptable general medical condition
11. Heterosexually active participants, male and female who are not surgically sterile or post-menopausal, must agree to use effective contraception, including abstinence, for the duration of the study and for 3 months after the study is completed
12. Have suitable facet joint anatomy for intra-articular injection
13. Willing and able to return for the follow-up (FU) visits
14. Able to read and understand study instructions, and willing and able to comply with all study procedures

Exclusion Criteria:

Participants must NOT meet any of the following exclusion criteria:

1. Hypersensitivity, allergy, or significant reaction to lidocaine or any ingredient of the study drug, including double-stranded DNA, mannose, and sucrose
2. Facet injection with corticosteroid in the past 6 months
3. Lumbar medial branch nerve ablation (e.g., by radiofrequency technique) within the past 12 months
4. Prior lumbar fusion surgery
5. Prior or existing medial branch nerve stimulation device (e.g., Mainstay device)
6. Scheduled surgical procedure or nerve ablation to joint within the next 6 months; participant agrees not to schedule a surgical procedure, nerve ablation, or added facet injection within 6 months of study treatment
7. High peri-operative risks which in the judgment of the investigator preclude a safe facet joint injection procedure (e.g. extreme obesity putting injection accuracy at risk, etc.)
8. Current treatment with immunosuppressive (systemic corticosteroid therapy [equivalent to >10 milligrams per day {mg/day} prednisone] or other strong immunosuppressant)
9. History of immunosuppressive therapy; high-potency systemic steroids in the last 3 months.
10. Currently receiving systemic chemotherapy or radiation therapy for malignancy
11. Clinically significant hepatic disease as indicated by clinical laboratory results ≥3 times the upper limit of normal for any liver function test (e.g., aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase)
12. Severe anemia (Grade 3; hemoglobin <8.0 grams per deciliter [g/dL], <4.9 millimoles per liter [mmol/L], <80 g/L; transfusion indicated), Grade 1 white cell counts (lymphocytes <Lower limit of normal [LLN] - 800/cubic millimeters [mm^3]; <LLN - 0.8 x 10^9/L, neutrophils <LLN - 1500/mm^3; <LLN - 1.5 x 10^9/L)
13. Positive serology with reflex for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus within 4 weeks of commencing the study
14. Significant neuropsychiatric conditions, dementia, major depression, or altered mental state that in the opinion of the Investigator will interfere with study participation
15. Current treatment with systemic antibiotics or antivirals (EXCEPTION: topical treatments)
16. Current treatment with anticoagulants, other than low-dose aspirin. Participants, if medically feasible, can interrupt anticoagulant therapy by following local medical practice protocol for intra-articular injections for participants on anticoagulant, antiplatelet therapy.
17. Known or suspected history of active alcohol or intravenous/oral drug abuse within 1 year before the screening visit
18. Use of any investigational drug or device within 1 month before enrollment or current participation in a trial that included intervention with a drug or device; or currently participating in an investigational drug or device study.
19. Any condition that, in the opinion of the Principal Investigator, could compromise the safety of the participant, the participant's ability to communicate with the study staff, or the quality of the data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Stokes, Study Director — Xalud Therapeutics; Howard Rutman, MD, Study Director — Xalud Therapeutics
Locations (3):
- United States (3):
  - Neurovations, Napa, California
  - Source HealthCare, Santa Monica, California
  - Center for Clinical Research, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo
Started | 25 | 25 | 25
Completed | 18 | 22 | 24
Not Completed | 7 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.71) | 58.0 (13.11) | 63.6 (13.74) | 60.3 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 13 | 34
  Male | 12 | 17 | 12 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 6
  Not Hispanic or Latino | 25 | 22 | 22 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 11
  White | 19 | 21 | 19 | 59
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.0 (6.23) | 31.0 (6.77) | 27.7 (6.44) | 29.9 (6.59)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) and Non-SAEs
Description: Adverse events were collected from the time of informed consent through the last study visit on Day 270 (9 months). Treatment Emergent Adverse Events (TEAEs) occurred from the time of study drug treatment on Day 0 through end of study (Day 270) or early termination.
Time Frame: Up to Day 270
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo
Number analyzed (Participants) | 25 | 25 | 25
Participants
  Any TEAEs: Yes | 11 | 12 | 14
  Any TEAEs: No | 14 | 13 | 11
  Related TEAEs: Yes | 1 | 1 | 3
  Related TEAEs: No | 24 | 24 | 22
  Serious TEAEs: Yes | 1 | 1 | 0
  Serious TEAEs: No | 24 | 24 | 25
  Related Serious TEAEs: Yes | 0 | 0 | 0
  Related Serious TEAEs: No | 25 | 25 | 25

2. Primary Outcome: Number of Participants Reporting Abnormal Hematology and Chemistry Parameters, Physical Examination, and Vital Signs
Description: Hematology and chemistry samples were only collected at Screening and not retested; therefore no results are available for those assessments Abnormal clinically significant physical examination findings were reported as adverse events, as applicable, and not separately reported.
  Vital signs of temperature, heart rate, respiratory rate and blood pressure were collected at all visits throughout the study.
Time Frame: Up to Day 270
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo
Number analyzed (Participants) | 25 | 25 | 25
Participants
  Day 0: Normal | 22 | 24 | 23
  Day 0: Abnormal - Not Clinically Significant | 3 | 1 | 2
  Day 0: Abnormal Clinically Significant | 0 | 0 | 0
  Day 0: Not Analyzed (Missing Data) | 0 | 0 | 0
  Day 270: Normal | 15 | 19 | 20
  Day 270: Abnormal - Not Clinically Significant | 0 | 1 | 0
  Day 270: Abnormal Clinically Significant | 0 | 0 | 0
  Day 270: Not Analyzed (Missing Data) | 10 | 5 | 5

3. Primary Outcome: Change From Baseline in Pain Intensity Using 0-100 Visual Analog Scale (VAS)
Description: The VAS is 0-100 scale which will be administered to participants via Electronic Patient Reported Outcome (ePRO) at each study visit. The participant will record his/her facet pain level on a scale from 0 (no pain) to 100 (worst pain). Higher scores indicate worse pain intensity.
Time Frame: Day 270
Population: Intent to Treat (ITT) population: All participants who were randomized who received the treatment injection analyzed according to randomized treatment. This was a phase 2a safety study that was not statistically powered for efficacy assessments.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo
Number analyzed (Participants) | 15 | 20 | 19
score on a scale | -38.12 (6.432) | -34.37 (5.717) | -42.32 (5.811)
Statistical Analysis 1: Comparison: 0.15mg XT-150 vs Placebo; This was a phase 2a safety study that was not statistically powered for efficacy assessments; Test type: Superiority; p = 1.00, Mixed Models Analysis; Mean Difference (Final Values) = 4.20, 95% CI 2-sided [-22.57 to 30.97], Standard Error of Mean 8.693
Statistical Analysis 2: Comparison: 0.45mg XT-150 vs Placebo; This was a phase 2a safety study that was not statistically powered for efficacy assessments; Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = 7.96, 95% CI 2-sided [-17.12 to 33.03], Standard Error of Mean 8.142

4. Secondary Outcome: Change From Baseline in Oswestry Disability Index (ODI) Scores
Description: The Oswestry Disability Index (ODI) is a 10-item questionnaire to quantify disability for acute or chronic low back pain. Each question is scored on a scale of 0 (least amount of disability) to 5 (most severe disability). Higher scores indicate severe disability.
Time Frame: Day 270
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo
Number analyzed (Participants) | 15 | 20 | 19
score on a scale | -14.4 (3.43) | -3.11 (3.104) | -8.25 (3.17)
Statistical Analysis 1: Comparison: 0.15mg XT-150 vs Placebo; This was a phase 2a safety study that was not statistically powered for efficacy assessments; Test type: Superiority; p = 0.1933, Mixed Models Analysis; Mean Difference (Final Values) = -6.15, 95% CI 2-sided [-15.49 to 3.19], Standard Error of Mean 4.676
Statistical Analysis 2: Comparison: 0.45mg XT-150 vs Placebo; This was a phase 2a safety study that was not statistically powered for efficacy assessments; Test type: Superiority; p = 0.2511, Mixed Models Analysis; Mean Difference (Final Values) = 5.14, 95% CI 2-sided [-3.73 to 14.00], Standard Error of Mean 4.434

5. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) Scores
Description: PGA is used to assess the current disease state on a 5-point Likert scale (1 = very good; 2 = good; 3 = fair; 4 = poor; and 5 = very poor). Higher score indicates worse symptoms.
Time Frame: Up to Day 270
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo
Number analyzed (Participants) | 15 | 20 | 19
score on a scale | -0.6 (1.55) | -0.7 (1.18) | -0.9 (0.97)

6. Secondary Outcome: Change From Baseline in International Physical Activity Questionnaire (IPAQ Short Form) Scores
Description: The globally standardized and validated IPAQ - short form is used to measure self-reported physical activity levels. Four metabolic equivalent tasks (MET) - vigorous, moderate, walking and sitting were included to obtain the physical activity levels from the participants. A higher MET value indicates a higher physical activity level.
Time Frame: Day 270
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo
Number analyzed (Participants) | 15 | 20 | 19
days
  Days vigorous physical activity during last 7 days | 0.7 (2.43) | -0.6 (1.64) | -0.3 (1.06)
  Days moderate physical activity during last 7 days | 1.5 (3.44) | -0.6 (3.45) | 0.2 (3.08)
  Days walking at least 10 minutes during last 7 days | 0.9 (2.64) | -0.8 (3.07) | -0.5 (3.27)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through the last study visit on Day 270 (9 months). Treatment Emergent Adverse Events occurred from the time of study drug treatment on Day 0 through end of study (Day 270) or early termination.
Arm/Group | 0.15mg XT-150 | 0.45mg XT-150 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 11/25 | 12/25 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.15mg XT-150 (N=25) | 0.45mg XT-150 (N=25) | Placebo (N=25)
Aortic Dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.15mg XT-150 (N=25) | 0.45mg XT-150 (N=25) | Placebo (N=25)
COVID-19 (Infections and infestations) | 5 | 1 | 4
Influenza (Infections and infestations) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is bound to terms and conditions of a Sponsored Clinical Trial Agreement which has strict confidentiality obligations running to Sponsor and broad provisions restricting PI's rights to publish or present any data or Study Results without Sponsor's express review consent and review.

DOCUMENTS (2):
  • Study Protocol (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT05196919/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT05196919/SAP_001.pdf